CLINICAL TRIAL: NCT00632554
Title: Phase 4, Randomized Study of Three Months-prednisolone Therapy in the Treatment of Chronic Eosinophilic Pneumonia
Brief Title: The Efficacy of Three Months-prednisolone Therapy for Chronic Eosinophilic Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Naoki Inui, Department of Respiratory Medicine, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hamamatsu-18-67
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Eosinophilic Pneumonia; Chronic Disease
MeSH Terms: conditions — Pulmonary Eosinophilia; Chronic Disease | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): prednisolone therapy for three months
  Interventions: Drug: prednisolone 0.5 mg/kg/day for three months
- 2 (Active Comparator): prednisolone therapy for six months
  Interventions: Drug: prednisolone 0.5 mg/kg/day for six months

INTERVENTIONS:
Drug: prednisolone 0.5 mg/kg/day for three months — period of treatment
  Other Names: prednisolone
  Arms: 1
Drug: prednisolone 0.5 mg/kg/day for six months — period of therapy
  Other Names: prednisolone
  Arms: 2

SUMMARY:
A comparison of 3 months-prednisolone administration with 6 months-prednisolone therapy in the treatment of chronic eosinophilic pneumonia. Three months-prednisolone administration may be as effective as 6 months-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven chronic eosinophilic pneumonia

Exclusion Criteria:

* Patients who received oral glucocorticosteroid (more than 10 mg)
* Immunosuppressive drug

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of 3 versus 6 months-prednisolone therapy for chronic eosinophilic pneumonia | Three years

SECONDARY OUTCOMES:
Safety of 3 versus 6 months-prednisolone therapy for chronic eosinophilic pneumonia | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Kingo Chida, MD, PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan

REFERENCES:
- [Derived] Oyama Y, Fujisawa T, Hashimoto D, Enomoto N, Nakamura Y, Inui N, Kuroishi S, Yokomura K, Toyoshima M, Yamada T, Shirai T, Masuda M, Yasuda K, Hayakawa H, Chida K, Suda T. Efficacy of short-term prednisolone treatment in patients with chronic eosinophilic pneumonia. Eur Respir J. 2015 Jun;45(6):1624-31. doi: 10.1183/09031936.00199614. Epub 2015 Jan 22. PMID 25614171